CLINICAL TRIAL: NCT05612477
Title: Blood Salvage in Orthotopic Liver Transplantation With HCC: A Randomized Open-labelled Trial of Effectiveness & Safety (SOLT Trial) - A Pilot Trial
Brief Title: Blood Salvage in Orthotopic Liver Transplantation With HCC
Acronym: SOLT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 20-5903
Record Dates: First submitted 2022-11-03; First posted 2022-11-10 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Hepatocellular Carcinoma; Surgery
Keywords: Liver transplantation
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Blood Transfusion, Autologous

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Autotransfusion (Experimental): patients in this arm will receive their salvaged and washed RBCs via transfusion
  Interventions: Procedure: Autotransfusion
- No Autotransfusion (No Intervention): patients in this arm will have their salvaged and washed RBCs discarded.

INTERVENTIONS:
Procedure: Autotransfusion — blood is collected from the surgical field, washed, processed and transfused back into the patient
  Arms: Autotransfusion

SUMMARY:
This single-centre randomized pilot study will investigate the feasibility, safety, and efficacy of IBSA (intraoperative blood cell salvage and autotransfusion -when a patient's own blood is collected from the surgical field, washed, and transfused back to them), in patients undergoing Liver transplantation for Hepatocellular carcinoma (HCC).

A total of 30 patient participants will be enrolled. A participant will be randomized only if enough blood is collected during the transplant surgery to produce a minimum of 1 unit of autologous blood. Patients will be randomized to receive their blood back (via transfusion) or have their own blood discarded. Patients will be followed after surgery for evaluation of safety and efficacy.

Depending on the outcomes of this feasibility trial, a subsequent larger full-scale multi-institutional trial will be planned, which will be more appropriately powered to evaluate the true impact of IBSA on the use of allogeneic blood products and post-transplant HCC-specific outcomes.

DETAILED DESCRIPTION:
Blood loss during liver transplantation (LT) often necessitates transfusion. However, allogeneic blood transfusion (blood from a donor) has risks. For this reason, intraoperative blood cell salvage and autotransfusion (IBSA) is frequently deployed to reduce the need for allogeneic blood transfusion. While IBSA is often used in LT, it is rarely used in patients undergoing LT for hepatocellular carcinoma (HCC) due to the theoretical risk of re-infusing cancer cells.

This single-centre, randomized, pilot study, will investigate the feasibility, safety, and efficacy of IBSA in patients undergoing LT for HCC.

Patients with HCC, listed for a Liver Transplant at the study institution, will be consented in clinic. At the time of liver transplant surgery, patients will be randomized, provided that enough blood is collected to generate a minimum of 1 unit of washed RBCs to give back. Participants randomized to arm 1 will receive their autologous blood via transfusion. Participants randomized to arm 2 will not receive their autologous blood - instead the blood will be discarded. Following surgery, participants will be followed for evaluation of safety and efficacy outcomes related to overall transfusions requirements and cancer recurrence.

The primary outcome is an evaluation of how many patients who consent to the trial will experience enough blood loss during surgery to be randomizable according to the study design (producing a minimum of 1 unit of washed RBCs).

Secondary outcomes include: whether the study can meet its accrual and enrollment goals within the study period; a comparison of rates of patient survival and HCC recurrence between the study groups; a comparison of the patient characteristics of those randomized to those not randomized. Blood will also be collected for correlative studies.

Depending on the outcomes of this feasibility trial, a subsequent larger full-scale multi-institutional trial will be planned, which will be more appropriately powered to evaluate the true impact of IBSA on the use of allogeneic blood products and post-transplant HCC-specific outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Listed for a liver transplant
* diagnosis of Hepatocellular carcinoma

Exclusion Criteria:

* - Patients with malignancy other than HCC, such as mixed cholangiocarcinoma-hepatocellular carcinoma, cholangiocarcinoma, and metastatic colorectal cancer. Patients who had a preoperative diagnosis of HCC but a postoperative diagnosis of any of the above will be analyzed separately.
* Pediatric patients (age<18 years at the time of screening)
* Patients undergoing re-transplantation
* Multi-organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-21 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility -Accrual | through study completion, an average of 24 months
  The primary outcome is an evaluation of how many patients who consent to the trial will experience enough blood loss during surgery to be randomizable according to the study design. This will be measured by comparing the number of consented patients undergoing LT who meet randomization requirements compared to those who do not.

SECONDARY OUTCOMES:
Feasibility- enrollment | 15 months
  to determine whether we can meet enrollment goals within the study period
Safety- HCC recurrence | 1 year post-transplant
  compare rates of HCC recurrence between groups

CONTACTS AND LOCATIONS:
Overall Officials: Gonzalo Sapisochin, MD, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada